CLINICAL TRIAL: NCT00759031
Title: Investigation of Dental Plaque and Gingival Index
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRO-2007-PLA-23-RR
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2008-11-25 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — fluorophosphate; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Marketed fluoride toothpaste (Placebo Comparator)
  Interventions: Drug: Sodium Monofluorophosphate
- B -Triclosan/NaF/CoPolymer toothpaste (Active Comparator)
  Interventions: Drug: Triclosan/Fluoride/Copolymer

INTERVENTIONS:
Drug: Sodium Monofluorophosphate — Brush teeth and evaluate plaque score after one use of the study toothpaste
  Other Names: Colgate Great Regular Flavor toothpaste
  Arms: A - Marketed fluoride toothpaste
Drug: Triclosan/Fluoride/Copolymer — Brush teeth and evaluate plaque score after one use of the study toothpaste
  Other Names: Colgate Total toothpaste
  Arms: B -Triclosan/NaF/CoPolymer toothpaste

SUMMARY:
Investigation of inhibitory effect of prototype toothpaste on dental plaque formation via modified gingival margin plaque index method.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 to 65 years inclusive
* Have a minimum of 20 natural uncrowned teeth (excluding 3rd molars) present
* Give written informed consent
* Be in good general health
* Must discontinue oral hygiene for 24-hrs.after initial appointment.
* No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredients in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

* Medical condition which requires pre-medication prior to dental visits/procedures
* Advanced periodontal disease
* 5 or more decayed, untreated dental sites
* Diseases of the soft or hard oral tissues
* Orthodontic appliances
* Abnormal salivary function
* Use of drugs that can currently affect salivary flow
* Use of antibiotics one (1) month prior to or during this study
* Use of any over the counter medications other than analgesics (i.e. aspirin, ibuprofen, acetaminophen, naproxyn)
* Pregnant or breastfeeding.
* Participation in another clinical study in the month preceding this study
* Allergic to common dentifrice ingredients.
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Corby, DDS, Principal Investigator
Locations (1):
- Boston University School of Dental Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Groups:
- Fluoride 1st, Triclosan +Fluoride 2nd: Subjects brushed their teeth once with Fluoride toothpaste and received plaque scores at baseline and 24 hours. After completed first intervention and washout, subjects used their second study treatment.
- Triclosan + Fluoride 1st, Fluoride 2nd: Subjects brushed their teeth once with the Triclosan + Fluoride toothpaste and then received plaque scores at baseline and 24 hours. After completed first intervention and washout, subjects used their second study treatment.
Period: First Intervention (1 Day)
Arm/Group | Fluoride 1st, Triclosan +Fluoride 2nd | Triclosan + Fluoride 1st, Fluoride 2nd
Started | 10 | 9
Completed | 8 | 8
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screening failure | 1 | 0
Period: Washout After 1st Intervention (1 Week)
Arm/Group | Fluoride 1st, Triclosan +Fluoride 2nd | Triclosan + Fluoride 1st, Fluoride 2nd
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Fluoride 1st, Triclosan +Fluoride 2nd | Triclosan + Fluoride 1st, Fluoride 2nd
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluoride 1st, Then Triclosan +Fluoride 2nd: Subjects brushed their teeth once with Fluoride toothpaste and received plaque scores at baseline and 24 hours. After completed first intervention and washout, subjects used their second study treatment.
- Triclosan + Fluoride 1st, Then Fluoride 2nd: Subjects brushed their teeth once with the Triclosan + Fluoride toothpaste and then received plaque scores at baseline and 24 hours. After completed first intervention and washout, subjects used their second study treatment.
- Total: Total of all reporting groups
Arm/Group | Fluoride 1st, Then Triclosan +Fluoride 2nd | Triclosan + Fluoride 1st, Then Fluoride 2nd | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.1 (11.14) | 33 (8.7) | 32.53 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Gingival Margin Plaque Index
Description: Scale 0 to 100% of tooth gingival margin covered by plaque. (0=no plaque, 100%=100% of the tooth's gingival margin is covered in plaque). The lower the score less dental plaque is present along the gum line and therefore the better the performance of the study treatment.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Fluoride: Subjects brushed their teeth once with Fluoride toothpaste and received plaque scores at baseline and 24 hours.
- Triclosan + Fluoride: Subjects brushed their teeth once with the Triclosan + Fluoride toothpaste and then received plaque scores at baseline and 24 hours.
Arm/Group | Fluoride | Triclosan + Fluoride
Number analyzed (Participants) | 16 | 16
Units on a scale | 15.4 (14.74) | 12.81 (14.06)
Statistical Analysis 1: Comparison: Fluoride vs Triclosan + Fluoride; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Fluoride | Triclosan + Fluoride
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days